CLINICAL TRIAL: NCT03280147
Title: Comparison of the Efficacy of a 7-day Versus 14-day Course of Intravenous Antibiotics in the Treatment of Uncomplicated Neonatal Bacterial Sepsis: a Randomized Controlled Non-inferiority Trial
Brief Title: 7 Days Versus 14 Days of Antibiotics for Neonatal Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Chacha Nehru Bal Chikitsalaya, New Delhi (Unknown); Lady Hardinge Medical College (Other Government); Indira Gandhi Institute of Child Health, Bangalore (Unknown); Institute of Obstetrics and Gynecology, Chennai (Unknown); King George's Medical University (Other); Pandit Bhagwat Dayal Sharma, PGIMS, Rohtak (Other); St Johns Medical College Hospital, Bangalore, India (Other)
Responsible Party: Principal Investigator, Sourabh Dutta, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5/7/329/2009-RHN
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Infant, Newborn; Neonatal SEPSIS; Anti-bacterial Agents; Recurrence
Keywords: Neonate; Sepsis; Antibiotics; Duration
MeSH Terms: conditions — Neonatal Sepsis; Recurrence; Sepsis

STUDY DESIGN:
Intervention Model Description: Randomized, outcome-assessor blinded, active-controlled, multi-centric, non-inferiority trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be provided objective clinical information related to episodes of all illnesses during follow-up with all patient identifiers removed and the record identified only by a unique code number. All imaging films and investigation reports provided to the outcome assessor will be similarly bereft of patient identifiers and coded by a unique code number. The outcome assessor will not be involved in the rest of the study. The outcome assessor will adjudicate whether the given episode of illness is a relapse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 7-day course of antibiotics (Experimental): Randomization of subjects will be performed at the end of 7 days of sensitive intravenous antibiotic administration, provided the subjects meet randomization criteria. Those who are randomized to the 7-day group will not receive any further antibiotics.
  Interventions: Drug: 7-day course of antibiotics
- 14-day course of antibiotics (Active Comparator): Randomization of subjects will be performed at the end of 7 days of sensitive intravenous antibiotic administration, provided the subjects meet randomization criteria. Those who are randomized to the 14-day group will receive 7 more days of the same antibiotics, to make it a total of 14 days.
  Interventions: Drug: 14-day course of antibiotics

INTERVENTIONS:
Drug: 7-day course of antibiotics — Subjects in the "7-day course of antibiotics" arm of the study will receive no further antibiotics after randomization as they would have already received 7 days of sensitive antibiotics before randomization. The choice of antibiotics would be guided by the blood culture and sensitivity report. Thus, subjects in this arm of the study could get a variety of antibiotics, depending on the sensitivity reports. Hence, names of specific antibiotics and/or their brand names have not been mentioned.
  Arms: 7-day course of antibiotics
Drug: 14-day course of antibiotics — Subjects in the "14-day course of antibiotics" arm of the study will receive 7 more days of antibiotics after randomization as they would have already received 7 days of sensitive antibiotics before randomization. The choice of antibiotics would be guided by the blood culture and sensitivity report. Thus, subjects in this arm of the study could get a variety of antibiotics, depending on the sensitivity reports. Hence, names of specific antibiotics and/or their brand names have not been mentioned.
  Arms: 14-day course of antibiotics

SUMMARY:
The optimum duration of intravenous antibiotic therapy for culture-proven neonatal bacterial sepsis is not known. Current practices, ranging from 7 days to 14 days of antibiotics, are not evidence-based. This is a randomized, active -controlled, multi-centric, non-inferiority trial to compare the efficacy of a 7-day course of intravenous antibiotics versus a 14-day course among neonates weighing > 1000 g at birth with culture-proven bacterial sepsis that is uncomplicated by meningitis, bone or joint infections deep-seated abscesses. The primary outcome measure is a definite or probable relapse within 21 days after stoppage of antibiotics.

DETAILED DESCRIPTION:
The optimum duration of intravenous antibiotic therapy for uncomplicated neonatal bacterial septicemia is not known. Pediatricians administer anywhere between 7 to 14 days of antibiotics, but these practices are not evidence based. C reactive protein (CRP) guided antibiotic duration is based on limited data and serial quantitative CRP is both cumbersome and not universally available. If it could be demonstrated that a 7-day course of antibiotics is not inferior to a 14-day course of antibiotics in terms of relapse rates of infection, then a 7 day course of antibiotics could be uniformly adopted, resulting in economic savings, shorter duration of hospitalization, less chances of hospital acquired infections, less chances of antibiotic induced adverse events and less antibiotic resistance. To test this hypothesis, a randomized, active-controlled, multi-centric, non-inferiority trial to compare the efficacy of a 7-day course of intravenous antibiotics with a 14-day course has been planned. Subjects weighing more than 1000 g at birth with suspected sepsis will be enrolled and observed for a 7-day period to see if they meet eligibility criteria for randomization. Subjects will be randomized on the 7th day of antibiotics, if the initial blood culture grows a non-Staphylococcus aureus bacterial organism, if they have no meningitis, osteomyelitis, septic arthritis or deep seated abscess and if the sepsis goes into clinical remission by the 5th day and remains in remission up to the 7th day of sensitive antibiotics. Subjects in the 14-day group will receive 7 more days of antibiotics after randomization, whereas those in the 7-day group will receive no further antibiotics after randomization. Subjects will be followed up for a 35-day period after randomization. The key outcome will be treatment failure as measured by "definite or probable relapse" within a 21-day period after completion of antibiotic therapy. Secondary outcomes will include definite relapse within 21 and 28 days after antibiotic completion and within 28 and 35 days after randomization; and probable relapse at similar time points. Other secondary outcomes will include secondary infections and adverse events. A total sample size of 700 (350 in each arm) will be required to detect a non-inferiority margin of 7%, assumed event rate of 10%, with 90% power, one-sided alpha error of 5% and loss to follow-up of approximately 10%. Data safety monitoring board will monitor serious adverse events in the trial and will perform at 1/3rd and 2/3rd of expected recruitment. At the time of interim analysis, the DSMB will revisit the sample size of the study. O'Brien Fleming's stopping criteria will be used for the primary outcome while Pocock's stopping rule will be used for the serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the initial observation part of study preceding randomization

1. Neonates aged 0-28 days, either inborn or outborn, who are currently admitted in the Neonatal Unit of the centre.
2. Whose birth weight is greater than or equal to1000 grams (it should be reliably ascertained from records of a hospital)
3. Whose residence is within approximately 15 kms from the center, so that the infant can be brought back to the center for follow-up
4. Who have suspected septicemia for which a conventional or BACTEC/BACTALERT blood culture is sent and for which the treating physician decides to start antibiotics

Inclusion criteria for Randomization applicable after 7 days of therapy of above patients with sensitive antibiotics:

1. Positive blood culture other than Staphylococcus aureus
2. No signs and symptoms of sepsis from end of day 5 through end of day 7 of starting sensitive antibiotics

Exclusion Criteria:

Exclusion criteria for the initial observation part of study preceding randomization:

1. Central Nervous System infection (Central Nervous System infection (meningitis will be defined as CSF Cells >25 per uL with polys >60% OR [(CSF glucose <20 mg/dL OR CSF:blood* glu ratio <0.6) AND (CSF protein >150 mg/dL in term OR >180 mg/dL in preterm)]
2. Septic arthritis, osteomyelitis or deep-seated abscess as clinically judged by the treating team
3. Life threatening congenital malformations as judged by the principal investigator of the centre

Exclusion criteria for randomization applicable after 7 days of therapy of above patients with sensitive antibiotics:

1. Sterile blood culture
2. Suspected contaminants in blood culture.
3. Growth of Staphylococcus aureus in blood culture
4. Growth of fungal organism in blood culture
5. Diagnosis of meningitis, septic arthritis, osteomyelitis, abscess
6. Has not gone into remission on day 5 or have recurrence of symptoms from day 5 through day 7
7. If the empiric antibiotic is resistant but neonate has shown improvement of signs and symptoms of sepsis and there is ambiguity regarding in vivo sensitivity of antibiotic use

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Definite or probable relapse within 21 days post-antibiotic completion as per protocol | From 0-21 days after the end of the planned antibiotic therapy
  Among participants who adhered to study protocol- Definite relapse: Episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode, Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Definite or probable relapse within 21 days post-antibiotic completion as per intention to treat | From 0-21 days after the end of the planned antibiotic therapy
  Among all randomized patients- Definite relapse: Episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode, Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.

SECONDARY OUTCOMES:
Definite relapse within 21 days post-antibiotic completion, as per protocol | From 0-21 days after the end of the planned antibiotic therapy
  Among participants who adhered to study protocol Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Definite relapse within 21 days post-antibiotic completion, as per intention-to-treat | From 0-21 days after the end of the planned antibiotic therapy
  Among all randomized patients Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Definite relapse within 28 days post-antibiotic completion, as per protocol | From 0-28 days after the end of the planned antibiotic therapy
  Among participants who adhered to study protocol Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Definite relapse within 28 days post-antibiotic completion, as per intention-to-treat | From 0-28 days after the end of the planned antibiotic therapy
  Among all randomized patients Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Definite relapse within 28 days post-randomization, as per protocol | From 0-28 days after randomization
  Among participants who adhered to study protocol Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Definite relapse within 28 days post-randomization, as per Intention-to-treat | From 0-28 days after randomization
  Among all randomized patients Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Definite relapse within 35 days post-randomization, as per protocol | From 0-35 days after randomization
  Among participants who adhered to study protocol Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Definite relapse within 35 days post-randomization, as per intention to treat | From 0-35 days after randomization
  Among all randomized patients Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode
Probable relapse within 21 days post-antibiotic completion, as per protocol | From 0-21 days after the end of the planned antibiotic therapy
  Among participants who adhered to study protocol Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Probable relapse within 21 days post-antibiotic completion, as per intention-to-treat | From 0-21 days after the end of the planned antibiotic therapy
  Among all randomized patients Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Probable relapse within 28 days post-antibiotic completion, as per protocol | From 0-28 days after the end of the planned antibiotic therapy
  Among participants who adhered to study protocol Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Probable relapse within 28 days post-antibiotic completion, as per intention-to-treat | From 0-28 days after the end of the planned antibiotic therapy
  Among all randomized patients Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Probable relapse within 28 days post-randomization, as per protocol | From 0-28 days after randomization
  Among participants who adhered to study protocol Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Probable relapse within 28 days post-randomization, as per intention-to-treat | From 0-28 days after randomization
  Among all randomized patients Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Probable relapse within 35 days post-randomization, as per protocol | From 0-35 days after randomization
  Among participants who adhered to study protocol Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Probable relapse within 35 days post-randomization, as per intention-to-treat | From 0-35 days after randomization
  Among all randomised patients Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Definite relapse or probable relapse within 28 days post-randomization, as per protocol | From 0-28 days after randomization
  Among participants who adhered to study protocol Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Definite relapse or probable relapse within 28 days post-randomization, as per Intention-to-treat | From 0-28 days after randomization
  Among all randomized patients Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Definite relapse or probable relapse within 35 days post-randomization, as per protocol | From 0-35 days after randomization
  Among participants who adhered to study protocol Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Definite relapse or probable relapse within 35 days post-randomization, as per intention-to-treat | From 0-35 days after randomization
  Among all randomised patients Definite relapse defined as: episode of blood-culture-positive relapse of neonatal sepsis caused by the same organism having the same antibiogram as the original episode Probable relapse: episode of illness without positive cultures adjudicated by a blinded adjudicator to be a relapse of the original episode of sepsis.
Secondary sepsis | From 0-35 days after randomization
  Sepsis due to bacterial organisms other than the original etiologic bacteria or with a different antibiogram or with a fungal organism
Adverse events | From 0-35 days after randomization
  Adverse events as per a list of adverse events, graded as per severity, and defined a priori

CONTACTS AND LOCATIONS:
Overall Officials: Sourabh Dutta, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (7):
- India (7):
  - Pandit BD Sharma Postgraduate Institute of Medical Sciences, Rohtak, Haryana
  - Indira Gandhi Institute of Child Health, Bangalore, Karnataka
  - Madras Medical College (for Institute of Obstetrics and Gynaecology), Chennai, Tamil Nadu
  - King Georges Medical University, Lucknow, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Kalawati Saran Childrens Hospital and Lady Hardinge Medical College, New Delhi
  - Chacha Nehru Bal Chikitsalaya, New Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dutta S, Nangia S, Jajoo M, Sundaram M, Kumar M, Shivanna N, Gathwala G, Nesargi S, Jain S, Kumar P, Saili A, Karthik A, Tripathi S, Bandiya P, Dalal P, Ray P, Randhawa VS, Saigal K, Radhakrishnan D, Venkatesh V, Jagannatha B, Sharma M, Nagaraj S, Malik M, Dogra S, Mittal S, Saini A, Makkar N, Dhir M, Chandramohan A, Pragati RA, Srivastava T, Mukundan L, Benakappa N, Shukla A, Rasaily R. Seven-day versus 14-day antibiotic course for culture-proven neonatal sepsis: a multicentre randomised non-inferiority trial in a low and middle-income country. Arch Dis Child Fetal Neonatal Ed. 2025 Oct 17;110(6):586-594. doi: 10.1136/archdischild-2024-328232. PMID 40280737

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03280147/Prot_004.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03280147/SAP_005.pdf